CLINICAL TRIAL: NCT06181721
Title: Evaluating Glucose Control Using a Next Generation Automated Insulin Delivery Algorithm in Patients With Type 1 and Type 2 Diabetes
Acronym: Evolution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVOLUTION
Record Dates: First submitted 2023-11-14; First posted 2023-12-26 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 Diabetes T2D; Type 1 Diabetes T1D; Omnipod; Automated Insulin Delivery System
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A with Type 1 Diabetes (Experimental): Participants with Type 1 Diabetes
  Interventions: Device: Omnipod 5 Automated Glucose Control System
- Group B with Type 2 Diabetes (Experimental): Participants with Type 2 Diabetes
  Interventions: Device: Omnipod 5 Automated Glucose Control System

INTERVENTIONS:
Device: Omnipod 5 Automated Glucose Control System — The Omnipod 5 Automated Glucose Control System will provide automated insulin delivery

SUMMARY:
To assess the safety and effectiveness of a next-generation automated insulin delivery algorithm in participants aged 16+ years with type 1 or type 2 diabetes.

DETAILED DESCRIPTION:
This study is a single-arm, observational clinical study that will enroll a maximum of 72 participants.

Participants between the ages of 16+ years with type 1 or type 2 diabetes currently using an insulin pump or receiving basal and bolus multiple daily injections (MDI), with an A1C between 7.5-11.0% at screening, will be recruited for the study.

Two participant groups will be recruited and will participate in up to 4 Phases:

* Group A (Participants with type 1 diabetes) will participate in Phase 1, Phase 2, Phase 3, and Phase 4
* Group B (Participants with type 2 diabetes) will participate in Phase 1, and Phase 4

Phase 1 (Group A and B) will include:

• 14 days of Standard Therapy while using a blinded Dexcom G6 CGM in an outpatient setting

Phase 2 (Group A only) will include:

• 48 hours of using build 1b.x of the Omnipod 5 System in Manual Mode in an outpatient setting

Phase 3 (Group A only) will include:

• 3 day/2 night supervised hotel stay using build 1b.x of the Omnipod 5 System in Automated Mode while also participating in meal and exercise challenges at a defined target glucose setting of 5.6 mmol/L (100 mg/dL). During the first 24 hours, participants will be instructed to not bolus for meals. For the following 24 hours, participants will be instructed to bolus for meals. At least 2 meals each day must contain at least 60 grams of carbohydrates. In addition, each day participants will take part in 45 minutes of exercise.

Phase 4 (Group A and B) will include:

• A total of 6 weeks using the Omnipod 5 System in Automated Mode in an outpatient setting at a defined target glucose setting of 5.6 mmol/L (100 mg/dL). During weeks 1-3, participants will be instructed to bolus for meals. During weeks 4-6, participants will be instructed to not bolus for meals.

After completion of a minimum of 10 participants for Group A, Phase 3, the data will be analysed and must meet prespecified criteria for Group A to proceed to Phase 4 and Group B to proceed to Phase 1 followed by Phase 4.

If the prespecified criteria are not met, software changes will be made and Group A, Phase 3 may be repeated either with the same participants or additional participants that meet the study criteria. Iterations of Group A, Phase 3 may continue until prespecified criteria are met.

ELIGIBILITY:
Inclusion Criteria-

Participants must meet all the following criteria to be included in the study:

1. Age at time of consent 16+ years
2. Individuals must be diagnosed with type 1 diabetes based on investigator's clinical judgment for at least 1 year. Individuals diagnosed with type 2 diabetes must be on basal and bolus insulin therapy, with no specified duration.
3. A1C between 7.5-11.0% at screening
4. Currently using U-100 rapid-acting insulin analogs with insulin pump or receiving multiple daily injections suitable for conversion to pump therapy for at least 3 months prior to study start
5. Willing to use a Dexcom G6 CGM for the duration of the study
6. Willing to use the Omnipod® 5 Automated Insulin Delivery System during the study
7. Willing to perform all fingerstick BG testing with their personal blood glucose meter at the frequency specified in the study protocol or per investigator discretion
8. Willing to participate in at least 45 minutes of exercise and meal challenges during the 3 day hotel stay (Group A only)
9. Willing to use carbohydrate counting for determination of meal boluses
10. Willing and able to sign the Informed Consent Form (ICF) and/or has a parent/guardian willing and able to sign the ICF.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the study:

1. Any medical condition, such as untreated malignancy, unstable cardiac disease, unstable or end-stage renal failure, eating disorders, or other conditions which in the opinion of the investigator, would put the participant at an unacceptable safety risk
2. Blood disorder or dyscrasia within 3 months prior to screening, including the use of hydroxyurea, which in the investigator's opinion could interfere with determination of HbA1C.
3. History of severe hypoglycemia within the past 6 months
4. History of diabetic ketoacidosis or hyperglycemic hyperosmolar syndrome in the past 6 months, unrelated to an intercurrent illness or infusion set failure
5. History of moderate to severe preproliferative or proliferative retinopathy based on screening within the last 12 months.
6. Planning to start a non-insulin anti-diabetic medication during the study. If on non-insulin medication, dose must be stable in the previous 30 days.
7. Planning to start a weight-loss agent during the study. If on a weight-loss medication, dose must be stable in the previous 30 days.
8. Currently on a low carbohydrate diet of < 60 grams of carbohydrates per day
9. Pregnant, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable forms of contraception include abstinence, barrier methods such as condoms, hormonal contraceptives, intrauterine device, surgical sterilisation such as tubal ligation or hysterectomy, or vasectomised partner)
10. Dermatological conditions at the proposed sensor/pump wear sites that in the investigator's opinion could preclude ability to wear the Pod and/or the Dexcom sensor
11. Current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the previous 12 months.
12. Currently on systemic steroids or intends to receive systemic steroid treatment in the next 6 months, including stable treatment for adrenal insufficiency. Inhaled, ophthalmic, topical, joint injection, and other locally applied steroids are allowed.
13. Currently participating in another clinical study using an investigational drug or device
14. Recent (within the preceding 30 days) participation in a clinical study using an investigational drug
15. Unable to follow the clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Percentage of time in hypoglycemic range (defined as < 3.9 mmol/L (<70 mg/dL)) | At the end of Phase 3 and Phase 4 to compare to baseline values
  Glucose metric from CGM
Percentage of time in hyperglycemic range (defined as > 13.9 mmol/L (>250 mg/dL)) | measured during the 9 week study phase
  Glucose metric from CGM

SECONDARY OUTCOMES:
Mean glucose value of all participants | Measured during the 9 week study phase
  Glucose metric from study provided continuous glucose monitor (CGM)
Percentage of time < 3.0 mmol/L (<54 mg/dL) | Measured during the 9 week study phase
  Glucose metric from CGM
Percentage of time > 10.0 mmol/L (>180 mg/dL) | Measured during the 9 week study phase
  Glucose metric from CGM
Percentage of time > 16.7 mmol/L (>300 mg/dL) | Measured during the 9 week study phase
  Glucose metric from CGM
Percentage of time between 3.9-10.0 mmol/L (70-180 mg/dL) | Measured during the 9 week study phase
  Glucose metric from CGM
Standard deviation and coefficient of variation | Measured during the 9 week study phase
  Glucose metric from CGM measured glucose variability with the coefficient of variation (CV)
Average total daily insulin (TDI) | Measured during the 9 week study phase
  measure of insulin
Average TDI/kg | Measured during the 9 week study phase
  measure of insulin
Average number of manual boluses/day | Measured during the 9 week study phase
  count of average number of insulin boluses
Average dose of insulin delivered by manual bolus/day | Measured during the 9 week study phase
  measure of insulin
Average number of hypoglycemic treatments when CGM is less than 3.9mmol/L | Measured during the 9 week study phase
  Glucose metric from CGM

CONTACTS AND LOCATIONS:
Locations (1):
- University of Otago, Christchurch, New Zealand